CLINICAL TRIAL: NCT00988247
Title: A Randomized, Double-Blind, Placebo-Controlled, Parallel-Group, Phase 3 Clinical Study to Assess the Long-term Efficacy and Safety of BDP HFA Nasal Aerosol (320 mcg, Once Daily) in Adult and Adolescent Subjects (12 Years of Age and Older) With Perennial Allergic Rhinitis (PAR)
Brief Title: Long Term Safety and Efficacy Trial of Beclomethasone Dipropionate - Hydrofluoroalkane (BDP-HFA) 320 mcg in Allergic Rhinitis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Teva Branded Pharmaceutical Products R&D, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: BDP-AR-303
Record Dates: First submitted 2009-09-30; First posted 2009-10-02 (Estimated); Results first posted 2012-05-23 (Estimated); Last update posted 2021-12-03 (Actual); Status verified 2021-12

CONDITIONS: Rhinitis, Allergic, Perennial
Keywords: Rhinitis, Allergic, Perennial; BDP-HFA; Hay fever; Allergic rhinitis
MeSH Terms: conditions — Rhinitis, Allergic, Perennial; Rhinitis, Allergic, Seasonal; Rhinitis, Allergic | interventions — Beclomethasone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- BDP HFA 320 µg/day (Experimental): During the 30-week (or 52-week, depending upon investigator site) double-blind Treatment Period participants self-administered 4 actuations (two per nostril) of 80 µg BDP HFA once daily each morning.
  Interventions: Drug: Beclomethasone dipropionate
- Placebo (Placebo Comparator): During the 30-week (or 52-week, depending upon investigator site) double-blind Treatment Period participants self-administered four actuations (two per nostril) of placebo HFA once daily each morning.
  Interventions: Drug: Placebo Nasal Aerosol

INTERVENTIONS:
Drug: Beclomethasone dipropionate — Total daily dose of 320 micrograms per day of beclomethasone dipropionate (BDP) hydrofluoroalkane (HFA) applied as a nasal aerosol each morning for 30-weeks (or 52-weeks, depending upon investigator site).
  Other Names: QNASL(TM)
  Arms: BDP HFA 320 µg/day
Drug: Placebo Nasal Aerosol — Placebo nasal aerosol administered daily for 30-weeks (or 52-weeks, depending upon investigator site).
  Arms: Placebo

SUMMARY:
Subjects with perennial allergic rhinitis will be randomized to 320 mcg of beclomethasone dipropionate (BDP) using a hydrofluoroalkane (HFA) propellant or placebo as a nasal aerosol. The subjects will be followed for safety and efficacy for a period of 30 or 52 weeks. BDP HFA is a steroid which is currently FDA approved for the treatment of asthma. BDP-HFA should be safe and effective as a "dry" nasal aerosol which may be preferred by some patients.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subjects, 12 years of age or older as of the Screening Visit (SV)
* General good health, and free of any concomitant conditions or treatment that could interfere with study conduct, influence the interpretation of study observations/results, or put the subject at increased risk during the study
* A history of PAR to a relevant perennial allergen for a minimum of two years immediately preceding the study Screening Visit (SV). The PAR must have been of sufficient severity to have required treatment (either continuous or intermittent) in the past, and in the investigator's judgment is expected to require treatment throughout the entire study
* A demonstrated sensitivity to at least one allergen known to induce PAR through a standard skin prick test. A positive test is defined as a wheal diameter at least 3 mm larger than the diluent control wheal for the skin prick test. Documentation of a positive result 12 months prior to Screening Visit (SV) is acceptable
* Other criteria apply

Exclusion Criteria:

* History of physical findings of nasal pathology, including nasal polyps or other clinically significant respiratory tract malformations, recent nasal biopsy, nasal trauma, including nasal piercing, or surgery and atrophic rhinitis or rhinitis medicamentosa (all within the last 60 days prior to Screening Visit [SV])
* Participation in any investigational drug study within the 30 days preceding the Screening Visit (SV) or planned participation in another investigational drug study at any time during this study
* History of a respiratory infection or disorder (including, but not limited to bronchitis, pneumonia, chronic sinusitis, or influenza within the 14 days preceding the Screening Visit (SV) or development of a respiratory infection during the Run-In Period
* Active asthma requiring treatment with inhaled or systemic corticosteroids and/or routine use of β-agonists and any controller drugs (e.g., theophylline, leukotriene antagonists). History of intermittent use (less than or equal to 3 uses per week) of inhaled short acting beta-agonists prior to the Screening Visit (SV) is acceptable.
* Other criteria apply

Randomization Criteria

* Subject continues to be in general good health, meeting the selection criteria
* Subject has a minimum subject-reported reflective TNSS of an average of 5 (out of a possible 12) on the last 7 days during the Run-In Period
* The subject-reported scores for rhinorrhea or nasal congestion must be an average of 2 or greater during the last 7 days of the Run-In Period
* Each subject must have adequately completed the electronic AR Assessment Diary (failure is defined as missing the diary entry on more than 2 calendar days during the last 7 days of the Run-In Period)
* Other criteria apply

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 529 (Actual)
Dates: Start 2009-10-31 (Actual); Primary Completion 2011-02-28 (Actual); Study Completion 2011-02-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Teva Branded
Locations (34):
- United States (34):
  - Teva Clinical Sudy Site, Oxford, Alabama
  - Teva Clinical Study Site, Encinitas, California
  - Teva Clinical Study Site, Huntington Beach, California
  - Teva Clinical Study Site, San Diego, California
  - Teva Clinical Study Site, Stockton, California
  - Teva Clinical Study Site, Colorado Springs, Colorado
  - Teva Clinical Study Site, Atlanta, Georgia
  - Teva Clinical Study Site, Stockbridge, Georgia
  - Teva Clinical Study Site, Normal, Illinois
  - Teva Clinical Study Site, Lenexa, Kansas
  - Teva Clinical Study Site, Overland Park, Kansas
  - Teva Clinical Study Site, Metairie, Louisiana
  - Teva Clinical Study Site, Wheaton, Maryland
  - Teva Clinical Study Site, Ypsilanti, Michigan
  - Teva Clinical Study Site, Minneapolis, Minnesota
  - Teva Clinical Study Site, Plymouth, Minnesota
  - Teva Clinical Study Site, Bozeman, Montana
  - Teva Clinical Study Site, North Syracuse, New York
  - Teva Clinical Study Site, Rochester, New York
  - Teva Clinical Study Site, Rockville Centre, New York
  - Teva Clinical Study Site, High Point, North Carolina
  - Teva Clinical Study Site, Cincinnati, Ohio
  - Teva Clinical Study Site, Sylvania, Ohio
  - Teva Clinical Study Site, Eugene, Oregon
  - Teva Clinical Study Site, Bethlehem, Pennsylvania
  - Teva Clinical Study Site, Collegeville, Pennsylvania
  - Teva Clinical Study Site, Dallas, Texas
  - Teva Clinical Study Site, El Paso, Texas
  - Teva Clinical Study Site, Houston, Texas
  - Teva Clinical Study Site, Kerrville, Texas
  - Teva Clinical Study Site, San Antonio, Texas
  - Teva Clinical Study Site, Vancouver, Washington
  - Teva Clinical Study Site, Greenfield, Wisconsin
  - Teva Clinical Study Site, West Allis, Wisconsin

REFERENCES:
- [Result] Meltzer EO, Jacobs RL, LaForce CF, Kelley CL, Dunbar SA, Tantry SK. Safety and efficacy of once-daily treatment with beclomethasone dipropionate nasal aerosol in subjects with perennial allergic rhinitis. Allergy Asthma Proc. 2012 May-Jun;33(3):249-57. doi: 10.2500/aap.2012.33.3571. PMID 22737708
- [Result] Meltzer EO, Jacobs RL, LaForce CF, Dorinsky PM, Kelley L, Dunbar SA, Tantry SK. . BDP HFA Nasal Aerosol 320 µg Once Daily Is Safe and Effective in the Treatment of Nasal Symptoms Associated With Perennial Allergic Rhinitis. Ann Allergy Asthma Immunol 2011 (Supplement); 107(11):A118 - Poster presentation.
- [Result] Carr W, Meltzer EO, Finn A, Dorinsky PM, Kelley L, Dunbar SA, Tantry SK. Effective nasal symptom relief and improvement in health-related quality of life in subjects with perennial allergic rhinitis following 6-week once-daily treatment with beclomethasone dipropionate hydrofluoroalkane nasal aerosol. J Allergy Clin Immunol 2012 (Supplement); 129:AB188 - Poster presentation
- [Result] Gross GN, Settipane RA, Ford LB, Kelley L, Dunbar SA, Tantry SK, Dorinsky PM . Patient Satisfaction and Ease-of-Use of BDP HFA Nasal Aerosol Device in Subjects With Perennial Allergic Rhinitis. Ann Allergy Asthma Immunol 2011 (Supplement); 107(11):A119 - Poster presentation
- [Derived] Weinstein SF, Andrews CP, Shah SR, Chylack LT Jr, Tankelevich A, Ding Y, Tantry SK. Long-term efficacy and safety of once-daily treatment with beclomethasone dipropionate nasal aerosol. Allergy Asthma Proc. 2014 Jul-Aug;35(4):323-31. doi: 10.2500/aap.2014.35.3767. PMID 24992552

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 857 patients were screened and 775 patients were enrolled in the study and participated in the Run-in Period. Of the 775 enrolled patients, 529 were randomized to study treatment.
Pre-assignment Details: During the 7 to 21 day Run-in Period, participants self-administered a single-blind placebo nasal aerosol once daily in the morning and assessed and recorded their daily seasonal rhinitis symptoms to determine eligibility for randomization.
Groups:
- BDP HFA 320 µg/Day: During the 30-week (or 52-week, depending upon investigator site) double-blind Treatment Period participants self-administered 4 actuations (two per nostril) of 80 µg beclomethasone dipropionate (BDP) hydrofluoroalkane (HFA) once daily each morning.
Period: Overall Study
Arm/Group | BDP HFA 320 µg/Day | Placebo
Started | 418 | 111
Safety Population | 415 (Participants who received at least 1 dose of study drug) | 111 (Participants who received at least 1 dose of study drug)
Intent to Treat Population | 414 (Participants who received at least 1 dose of study drug and had at least 1 post-baseline assessment) | 110 (Participants who received at least 1 dose of study drug and had at least 1 post-baseline assessment)
Completed | 335 | 85
Not Completed | 83 | 26
Not completed — Adverse Event | 17 | 3
Not completed — Withdrawal by Subject | 44 | 13
Not completed — Pregnancy | 1 | 2
Not completed — Lost to Follow-up | 11 | 2
Not completed — Protocol Violation | 4 | 5
Not completed — Sponsor requested withdrawal | 3 | 1
Not completed — Other | 3 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | BDP HFA 320 µg/Day | Placebo | Total
Number analyzed (Participants) | 414 | 110 | 524
Age, Continuous [Mean (Standard Deviation); unit: years] — Demographic data are provided for the Intent to Treat population.
  years | 37.4 (13.6) | 35.7 (12.9) | 37.1 (13.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 286 | 66 | 352
  Male | 128 | 44 | 172
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 45 | 12 | 57
  Not Hispanic or Latino | 369 | 98 | 467
  Unknown or Not Reported | 0 | 0 | 0
Race/Ethnicity, Customized [Number; unit: participants] — A participant may select more than one race type.
  participants
    American Indian or Alaska Native | 7 | 2 | 9
    Asian | 13 | 1 | 14
    Native Hawaiian or Other Pacific Islander | 3 | 0 | 3
    Black or African American | 63 | 14 | 77
    White | 341 | 97 | 438
    Unknown or Not Reported | 1 | 0 | 1
Body mass index [Mean (Standard Deviation); unit: kg/m^2] | 28.8 (6.7) | 28.4 (6.7) | 28.7 (6.7)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Average Subject-Assessed 24-Hour Reflective Total Nasal Symptom Score (rTNSS) up to 30 Weeks
Description: Participants recorded the severity of their nasal symptoms (sneezing, runny nose, itchy nose and nasal congestion) in the past 24-hours (prior to the assessment) daily using the following scale:
  0=absent (no sign/symptom); 1=mild (sign/symptom present, easily tolerated); 2=moderate (bothersome but tolerable); 3=severe (hard to tolerate, interfere with daily activities).
  The total nasal symptom score (sum of 4 symptom scores) ranges from 0 to 12 (worst symptoms). A negative change from baseline score indicates improvement.
Time Frame: Baseline (Days -6 to 0), Day 1 to Week 30
Population: Intent to treat population
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | BDP HFA 320 µg/Day | Placebo
Number analyzed (Participants) | 414 | 110
units on a scale | -3.4 (0.11) | -2.4 (0.22)
Statistical Analysis 1: Comparison: BDP HFA 320 µg/Day vs Placebo; Test type: Superiority or Other; p < 0.001, ANCOVA; The repeated measures ANCOVA included covariate adjustment for baseline, treatment, week and the treatment by week interaction; LS mean treatment diff from placebo] = -0.97, 95% CI 2-sided [-1.5 to -0.5]

2. Secondary Outcome: Change From Baseline in Average Subject-Assessed 24-Hour Instantaneous Total Nasal Symptom Score (iTNSS) up to 30 Weeks
Description: Participants recorded the severity of their nasal symptoms (sneezing, runny nose, itchy nose and nasal congestion) in the past 10 minutes (prior to the assessment) daily using the following scale:
  0=absent (no sign/symptom); 1=mild (sign/symptom present, easily tolerated); 2=moderate (bothersome but tolerable); 3=severe (hard to tolerate, interfere with daily activities).
  The total nasal symptom score (sum of 4 symptom scores) ranges from 0 to 12 (worst symptoms). A negative change from baseline score indicates improvement.
Time Frame: Baseline (Days -6 to 0), Day 1 to Week 30
Population: Intent to treat population
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | BDP HFA 320 µg/Day | Placebo
Number analyzed (Participants) | 414 | 110
units on a scale | -2.9 (0.11) | -2.0 (0.21)
Statistical Analysis 1: Comparison: BDP HFA 320 µg/Day vs Placebo; Test type: Superiority or Other; p < 0.001, ANCOVA; [statistical method as in outcome 1, analysis 1]; LS mean treatment diff from placebo] = -0.96, 95% CI 2-sided [-1.4 to -0.5]

3. Secondary Outcome: Change From Baseline in Average Subject-Assessed 24-Hour Reflective Total Nasal Symptom Score (rTNSS) up to 52 Weeks
Description: as for outcome 1
Time Frame: Baseline (Days -6 to 0), Day 1 to Week 52
Population: Intent to treat population.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | BDP HFA 320 µg/Day | Placebo
Number analyzed (Participants) | 414 | 110
units on a scale | -3.7 (0.12) | -2.6 (0.23)
Statistical Analysis 1: Comparison: BDP HFA 320 µg/Day vs Placebo; Test type: Superiority or Other; p < 0.001, ANCOVA; [statistical method as in outcome 1, analysis 1]; LS mean treatment diff from placebo] = -1.09, 95% CI 2-sided [-1.6 to -0.6]

4. Secondary Outcome: Change From Baseline in Average Subject-Assessed 24-Hour Instantaneous Total Nasal Symptom Score (iTNSS) up to 52 Weeks
Description: as for outcome 2
Time Frame: Baseline (Days -6 to 0), Day 1 to Week 52
Population: Intent to treat population
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | BDP HFA 320 µg/Day | Placebo
Number analyzed (Participants) | 414 | 110
units on a scale | -3.1 (0.11) | -2.0 (0.22)
Statistical Analysis 1: Comparison: BDP HFA 320 µg/Day vs Placebo; Test type: Superiority or Other; p < 0.001, ANCOVA; [statistical method as in outcome 1, analysis 1]; LS mean treatment diff from placebo] = -1.10, 95% CI 2-sided [-1.6 to -0.6]

5. Secondary Outcome: Change From Baseline to Week 30 in Rhinoconjunctivitis Quality of Life Questionnaire (RQLQ) in Participants With Impaired Quality of Life at Baseline
Description: The adult RQLQ has 28 questions in 7 domains (activities, sleep, non-nose/eye symptoms, practical problems, nasal symptoms, eye symptoms, and emotional). Participants were asked to recall their experiences during the previous week and to give their responses on a 7-point scale (0 = Least severe to 6 = Extremely severe). The overall RQLQ score is the mean of all 28 responses, and ranges from 0 to 7.
  Week 30 scores were compared to baseline scores. A negative change score indicates improvement.
Time Frame: Day 0 (Baseline) and Week 30
Population: The RQLQ population included only those participants over the age of 18 years with an impaired quality of life at Baseline as defined by a RQLQ score at Day 0 of 3.0 or greater.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | BDP HFA 320 µg/Day | Placebo
Number analyzed (Participants) | 202 | 50
units on a scale | -2.2 (0.09) | -1.9 (0.19)
Statistical Analysis 1: Comparison: BDP HFA 320 µg/Day vs Placebo; Test type: Superiority or Other; p = 0.143, ANCOVA; ANCOVA with treatment, baseline and pooled center in the model; treatment difference = -0.30, 95% CI 2-sided [-0.7 to 0.1]

6. Secondary Outcome: Change From Baseline to Week 52 in Rhinoconjunctivitis Quality of Life Questionnaire (RQLQ) in Participants With Impaired Quality of Life at Baseline
Description: The adult RQLQ has 28 questions in 7 domains (activities, sleep, non-nose/eye symptoms, practical problems, nasal symptoms, eye symptoms, and emotional). Participants were asked to recall their experiences during the previous week and to give their responses on a 7-point scale (0 = Least severe to 6 = Extremely severe). The overall RQLQ score is the mean of all 28 responses, and ranges from 0 to 7.
  Week 52 scores were compared to baseline scores. A negative change score indicates improvement.
Time Frame: Day 0 (Baseline) and Week 52
Population: as for outcome 5
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | BDP HFA 320 µg/Day | Placebo
Number analyzed (Participants) | 109 | 23
units on a scale | -2.0 (0.14) | -1.5 (0.30)
Statistical Analysis 1: Comparison: BDP HFA 320 µg/Day vs Placebo; Test type: Superiority or Other; p = 0.130, ANCOVA; ANCOVA with treatment, baseline and pooled center in the model; treatment difference = -0.49, 95% CI 2-sided [-1.1 to 0.1]

ADVERSE EVENTS:
Arm/Group | BDP HFA 320 µg/Day | Placebo
Serious Adverse Events (participants affected / at risk) | 8/415 | 3/111
Other Adverse Events (participants affected / at risk) | 216/415 | 37/111
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | BDP HFA 320 µg/Day (N=415) | Placebo (N=111)
Nephrolithiasis (Renal and urinary disorders) | 1 | 0
Intraocular pressure increased (Investigations) | 1 | 0
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
Bladder injury (Injury, poisoning and procedural complications) | 1 | 0
Menorrhagia (Reproductive system and breast disorders) | 1 | 0
Pelvic adhesions (Reproductive system and breast disorders) | 1 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Fall (Injury, poisoning and procedural complications) | 1 | 0
Humerus fracture (Injury, poisoning and procedural complications) | 1 | 0
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 1 | 0
Ovarian cyst (Reproductive system and breast disorders) | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1
Viral infection (Infections and infestations) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | BDP HFA 320 µg/Day (N=415) | Placebo (N=111)
Nasopharyngitis (Infections and infestations) | 67 | 14
Sinusitis (Infections and infestations) | 34 | 8
Upper respiratory tract infection (Infections and infestations) | 43 | 7
Headache (Nervous system disorders) | 28 | 6
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 44 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor has the right 60 days before submission for publication to review/provide comments. If the Sponsor's review shows that potentially patentable subject matter would be disclosed, publication or public disclosure shall be delayed for up to 90 additional days in order for the Sponsor, or Sponsor's designees, to file the necessary patent applications. In multicenter trials, each PI will postpone single center publications until after disclosure or publication of multicenter data.